CLINICAL TRIAL: NCT04268043
Title: Comparation of Efficacy and Safety of Proseal Laryngeal Mask Airway With Flexible Laryngeal Airway Mask in Otitis Media Surgery
Brief Title: Comparation of Proseal Laryngeal Mask Airway With Flexible Laryngeal Airway Mask
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2019041-2
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia Intubation Complication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flexible laryngeal airway (Experimental)
  Interventions: Device: flexible laryngeal airway mask
- proseal laryngeal mask airway (Experimental)
  Interventions: Device: proseal laryngeal mask airway

INTERVENTIONS:
Device: flexible laryngeal airway mask — Ventilation with flexible laryngeal mask airway
  Arms: flexible laryngeal airway
Device: proseal laryngeal mask airway — Ventilation with proseal laryngeal mask airway
  Arms: proseal laryngeal mask airway

SUMMARY:
Objective To investigate the comparative effect of proseal laryngeal mask airway and flexible laryngeal airway mask during otitis media surgery. Methods 200 patients of ASA I or II classification, 18-65 years old, BMI<30 kg/m2 undergoing otitis media surgery are randomly divided into two groups (Group P with proseal laryngeal mask airway and Group F with flexible laryngeal airway mask, respectively). After induction, selecting a appropriate size of LMA to patient,s weight, using the standard index finger-guided technique inserting the LMA, and then the patients were ventilated mechanically. The success rate of inserting laryngeal mask, the intubation time, surgery time and wake time were also recorded. Tidal volume and leakage pressure in patients with supine and lateral positioning were assessed respectively. The scale of fiberoptic bronchoscopy was also recorded to show airway exposure. Related complications such as sore throat, hoarseness, cough, laryngospasm, bloating, nausea and vomiting, soft tissue injury, blood residue after pulling out the LMA were analyzed.Postoperative voice and laryngopharyngeal symptom are also recorded.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of otitis media.

Exclusion Criteria:

Problems with the upper airway. Gastric carcinoma. Reflux esophagitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
successful insert rate | 0 minute after insertion
  success rate of inserting laryngeal mask
tidal volume | 5 minute afer successful insertion
  tidal volume at 15cmH2O in patients with supine and lateral positioning
leakage pressure | 5 minute afer successful insertion
  leakage pressure in patients with supine and lateral positioning
The scale of fiberoptic bronchoscopy | 0 minute afer successful insertion
  1 = only vocal cords visible; 2 = vocal cords plus posterior epiglottis visible; 3 = vocal cords plus anterior epiglottis visible; and 4 = vocal cords invisible
Number of Participants with cranial nerve injury | 1hours after the surgery
  Number of Participants with cranial nerve injury

SECONDARY OUTCOMES:
Number of Participants with sore throat | 1hours after the surgery
  Number of Participants with sore throat
Number of Participants with hoarseness | 1hours after the surgery
  Number of Participants with hoarseness
Number of Participants with cough | 1hours after the surgery
  Number of Participants with cough
Number of Participants with laryngospasm | 1hours after the surgery
  Number of Participants with laryngospasm
Number of Participants with soft tissue injury | 1hours after the surgery
  Number of Participants with soft tissue injury